CLINICAL TRIAL: NCT00782041
Title: Phase II Study of Oxaliplatin in Combination With 5-fluorouracil (5-FU) and Folinic Acid (FA) in Patients Who Have Failed First-line Treatment for Locally Advanced or Metastatic Cervical Cancer.
Brief Title: Patients Who Have Failed First Line Treatment for Locally Advanced and/or Metastatic Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: protocol violation
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8311
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Uterine Neoplasms
MeSH Terms: conditions — Uterine Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Oxaliplatin 85 mg/m² over 3 hours at Day 1 and Day 15. 5-FU 2,000 mg/m² over 4 hours at Day 1. Folinic acid 20 mg/m² Bolus at Day 1.
  Interventions: Drug: Oxaliplatin; Drug: 5-FluoroUracil; Drug: Folinic acid

INTERVENTIONS:
Drug: Oxaliplatin — 85 mg/m²
Drug: 5-FluoroUracil — 2,000 mg/m²
Drug: Folinic acid — 20 mg/m²

SUMMARY:
Primary:

* To assess the overall response rate of oxaliplatin in patients with bidimensionally measurable disease at baseline.

Secondary:

* To assess the safety and tolerability of oxaliplatin
* To assess time to progression and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Have Locally advanced/metastatic squamous or adenocarcinoma of the cervix
* Prior therapy with cisplatin allowed
* First-line treatment may have been surgery,radiotherapy or chemotherapy either as a single agent or multi-modality therapy
* Must have measurable disease
* Histologically Proven Carcinoma of the cervix
* ECOG PS ≤2
* No other serious concomitant illness
* Fully recovered from any prior therapy
* Lab: ANC >1500 mm³, Platelets > 100000 mm³, Creatinine ≤ 1.5 x Normal value, Bilirubin ≤ 1.5 x Normal value, SGPT (ALT) ≤ 2.5 x Normal value

Exclusion Criteria:

* Known allergy to one of the study drugs
* Peripheral neuropathy > grade2

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-01; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Response rate | Throughout the study period

SECONDARY OUTCOMES:
Progression-free survival | Throughout the study period
Overall survival | Throughout the study period
Adverse events | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Paibulsirijit Sompob, MD, Study Director — Sanofi
Locations (1):
- Sanofi aventis administrative office, Bangkok, Thailand